CLINICAL TRIAL: NCT00426465
Title: Neural Substrates of Lasting Motor Skill Learning by Spacing Effect
Brief Title: Spaced Versus Massed Skill Learning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070072; 07-N-0072
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-12-16

CONDITIONS: Healthy Volunteer
Keywords: Motor Practice; Magnetic Stimulation; Stroke; Spacing Effect; Massed Practice; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
This study will explore the optimum training schedule for stroke patients to learn motor skills. It will see if motor training is more effective when training sessions are distributed over time (spaced training) or when the sessions are scheduled close together (massed training). The results of this study may help researchers devise the best training schedule for patients to derive the maximum benefit from rehabilitation therapy.

Healthy normal volunteers and people who have had a stroke may be eligible for this study. Patients must be 3 months post-stroke. All participants must be right-handed and between 18 and 80 years of age.

Participants practice a pinch motor task and receive transcranial magnetic stimulation (TMS). Hand muscle activity is measured using surface electromyography (EMG). Pinch training involves training the participant to pinch as strongly as possible, using a device that records the force. For TMS, a wire coil is held on the subject s scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg. For surface EMG, electrodes (small metal disks) are filled with a conductive gel and taped to the skin over the muscle.

Following one practice session of pinch task training and TMS, participants have four training sessions, which are scheduled 24 hours, 2 weeks, 1 month and 3 months after the practice session.

For the 4- to 5-hour practice session, subjects do the following:

* Perform a single session of pinch motor task for familiarization
* Undergo TMS to measure brain activity
* Practice five 6-minute blocks of pinch motor task with rest periods between sessions and perform a calculation task (addition and subtraction tasks) during each rest period
* Receive TMS over 15 minutes. (Some sessions may have sham TMS.)
* Read books and magazines during a 45-minute rest period
* Perform a single block of the pinch motor task
* Undergo TMS to measure brain activity
* Complete a questionnaire that measures attention, fatigue and mood

For the remaining four sessions, participants perform one practice block and TMS. Each session lasts about 2 hours.

DETAILED DESCRIPTION:
In cognitive psychology, practice is most effective when training sessions are distributed over time (spaced), rather than when they are close to each other (massed). This phenomenon, thought to engage long-term potentiation-like mechanisms in animal models and described as spacing effect, has not been investigated in the motor domain. It is not known if spaced motor training elicits longer lasting learning effects than massed motor training.

Objective and Study Population:

The purpose of this investigation is to assess the relevance of the spacing effect in motor skill learning in healthy volunteers and in patients with chronic stroke.

Design:

Experiment 1: Determination of long term learning in healthy volunteers with spaced and massed practice:

The first hypothesis is that spaced practice will enhance long-lasting learning of a motor task (defined as performance improvements measured 1 and 3 months post training) to a larger extent than massed practice in separate groups of healthy volunteers. Healthy volunteers will practice a well-characterized pinch force task following spaced or massed schedules in a factorial design (n=26). If this hypothesis is proven correct, we will proceed as suggested by PIRC, to Experiments 2 and 3, to gain information on the mechanisms underlying the superior training strategy in healthy volunteers (Exp 2) and to determine if this training strategy is also superior to massed practice in stroke patients (Exp 3), an issue of crucial importance in neurorehabilitation.

Experiment 2: Study of mechanisms underlying superior effects of spaced over massed practice in healthy volunteers, rTMS:

Previous work demonstrated the involvement of the primary motor cortex (M1) in consolidation of motor learning and the importance of top-down attentional control by the prefrontal cortex. It is possible that an enhanced recruitment of these two regions mediates the superior performance levels reached with spaced training. Here, we plan to study the effects of inhibitory 1 Hz TMS applied to M1 and PFC on performance improvements with spaced training. We hypothesize that the superiority of spaced practice, relative to massed practice, will be cancelled by down regulation of activity in M1 and PFC but not by sham or posterior parietal cortex (PPC) stimulation (n=104).

Experiment 3: Determination of long term learning in stroke patients with spaced and massed practice:

We hypothesize that motor learning in chronic stroke patients will improve to a larger extent with spaced than with massed practice (n=42).

This study is expected to delineate the role of the spacing effect on human motor learning and identify two of the possible neural cortical substrates in healthy volunteers and its possible beneficial effects on motor learning after stroke.

Experiment 4: Determination of whether original findings with the spacing effect in explicit motor learning generalized to implicit/procedural motor learning:

The ability to generalize to implicit motor learning is important because implicit learning (also known as procedural learning), which is defined as learning which occurs without awareness and without intention, underlies the development of automaticity which characterizes all well-learned motor skills (Reber, 1993; Squire, 2004). Hence, for the purposes of stroke rehabilitation, it is important to determine if and how the spacing effect occurs for implicit (procedural) learning which underlies the development of automaticity that characterizes all well-learned motor skills. In addition, using explicit motor sequencing tasks, it is difficult to determine if the spacing effect helps general motor skill or sequence-specific skill. In other words, performance benefits from the spacing effect can derive from improvements in the visuomotor transformation required to push the keys on the board independently of the presence or absence of sequence, or from motor sequencing improvements. Both of these issues can be addressed using the serial reaction time task (or SRTT), a well-studied implicit motor sequence learning task which is described in more detail in this protocol (Nissen and Bullemer, 1984).

We hypothesize that the spacing effect occurs in a sequence-specific manner for implicit motor sequence learning. We hypothesize that an SMA-based motor network underlies the superiority of the spacing effect for implicit motor sequence learning. We will show this by using 1Hz TMS to create virtual lesions and establish a cause-effect link between the SMA (or M1 but not CZ or sham) and superior motor skill with Spaced over Massed training (n=80).

Outcome Measures:

The primary outcome measure will be improvement in pinch force. Secondary outcome measurements will be measures of motor cortical excitability including motor evoked potential amplitudes, intracortical inhibition and facilitation.

For procedural/implicit motor sequence learning, the primary outcome measure will be an improvement in skill as seen by a difference in reaction time between sequenced and randomly ordered trials.

ELIGIBILITY:
* INCLUSION CRITERIA: Healthy Volunteers
* Age between 18-80 years
* Able to perform tasks required by the study<TAB>
* Willing and able to give consent
* Have a normal physical and neurological examination
* Right Handed as assessed by the Edinburgh inventory scale (Edinburgh, 1971)

EXCLUSION CRITERIA: Healthy Volunteers

* History of alcohol or drug abuse, and psychiatric illness such as severe depression.
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.

INCLUSION AND EXCLUSION CRITERIA FOR STROKE PATIENTS:

Patients must be between the ages of 18 and 80 years of age, inclusive. Included will be those with chronic (more than 3 months) stroke who recovered motor function to the point of being able to perform the ballistic pinch force task. Stroke patients will be recruited through the NIH Clinical Research Volunteer Program. Assessment of severity of initial hemiparesis will be taken either from patient report or medical records.

EXCLUDED FROM THE STUDY WILL BE PATIENTS:

1. with a history of severe alcohol or drug abuse, psychiatric illness like severe depression, severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam (Folstein, 1976) score of 23 or less)
2. with severe uncontrolled medical problems (e.g., cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others)
3. with metal in the body (metal in the cranium, metal fragments from occupational exposure, surgical clips in or near the brain, cardiac or neural pacemakers, intracardiac lines, implanted medication pumps, blood vessel, cochlear or eye implants)
4. with history of loss of consciousness or epilepsy
5. with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2007-01-17; Study Completion 2013-12-16

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bermpohl F, Fregni F, Boggio PS, Thut G, Northoff G, Otachi PT, Rigonatti SP, Marcolin MA, Pascual-Leone A. Left prefrontal repetitive transcranial magnetic stimulation impairs performance in affective go/no-go task. Neuroreport. 2005 Apr 25;16(6):615-9. doi: 10.1097/00001756-200504250-00020. PMID 15812319
- [Background] Bermpohl F, Fregni F, Boggio PS, Thut G, Northoff G, Otachi PT, Rigonatti SP, Marcolin MA, Pascual-Leone A. Effect of low-frequency transcranial magnetic stimulation on an affective go/no-go task in patients with major depression: role of stimulation site and depression severity. Psychiatry Res. 2006 Jan 30;141(1):1-13. doi: 10.1016/j.psychres.2005.07.018. Epub 2005 Dec 13. PMID 16352348
- [Background] Bridgers SL, Delaney RC. Transcranial magnetic stimulation: an assessment of cognitive and other cerebral effects. Neurology. 1989 Mar;39(3):417-9. doi: 10.1212/wnl.39.3.417. PMID 2927652